CLINICAL TRIAL: NCT02079974
Title: Statins: A New Therapeutic Option for Treatment of Patients With Endometriosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Robert F. Casper (Other)
Responsible Party: Sponsor-Investigator, Dr. Robert F. Casper, Professor, Dept of Obstetrics and Gynecology, Toronto Centre for Advanced Reproductive Technology
Organization: Toronto Centre for Advanced Reproductive Technology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4169720110; NCT02084667 (obsolete NCT alias)
Record Dates: First submitted 2014-03-03; First posted 2014-03-06 (Estimated); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Endometriosis
Keywords: endometriosis; pain; fertility
MeSH Terms: conditions — Endometriosis; Pain | interventions — Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pravastatin (Experimental): Pravastatin sodium 20mg PO daily
  Interventions: Drug: Pravastatin

INTERVENTIONS:
Drug: Pravastatin — 20 mg pravastatin sodium daily for 3 months
  Other Names: pravastatin sodium

SUMMARY:
Endometriosis is a chronic inflammatory disorder leading to painful periods, pain with intercourse and infertility. The available treatment options to alleviate pain involve mainly hormonal treatments and surgery. All current hormonal treatments are effective but disrupt the normal variations in reproductive hormones which prevent ovulation, and thus pregnancy. Statins, a group of cholesterol lowering drugs, have anti-inflammatory properties which may be helpful also for the pain related to endometriosis. The investigators plan to undertake a pilot study of 10 patients with endometriosis who will take pravastatin sodium together with coQ10, which is inhibited by statins, for a period of 3 months. If this pilot study shows that the statin treatment may decrease pain symptoms in endometriosis, then the investigators plan to undertake a larger study to further investigate this matter.

DETAILED DESCRIPTION:
* Initial grading of pain by a Linear Analogue Scale (LAS) from 1-10
* Initial blood biochemistry including liver function test, lipid profile, creatine/BUN, creatine kinase
* 3 months of treatment with statins (Pravastatin) in a dose of 40mg daily
* Supplementation with CoQ10 (200mg) daily for 3 months

ELIGIBILITY:
Inclusion Criteria:

* female patients of reproductive age group (18-38 years) with a clinical or surgical diagnosis of endometriosis with pain symptoms

Exclusion Criteria:

* use of hormonal suppression for pain control (OCP, GnRHa) within 6-months
* history of surgery for endometriosis within 6- months
* current renal or hepatic active disease
* current or history of myopathic disease
* medication that may interact with statins (erythromycin, gemfibrosil, antifungals, antiretrovirals, other cholesterol lowering drugs)

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
subjective assessment of pain | 3 months
  Linear analogue scale for each component of pain (dysmenorrhea; pelvic pain; dyspareunia)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Casper, MD, Principal Investigator — Dept of Obstetrics and Gynecology, University of Toronto
Locations (1):
- Mount Sinai Hospital, University of Toronto, Toronto, Ontario, Canada